CLINICAL TRIAL: NCT05558137
Title: An Observational Study of Mivacurium 0.2 mg/kg, Comparing Onset Time, Duration of Action and Effect on Intubating Conditions in Young (18 - 40 Years) and Elderly (= 80 Years) Patients
Brief Title: Mivacurium 0.2 mg/kg in Young (18 - 40 Years) and Elderly (= 80 Years) Patients
Status: Completed | Type: Observational
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-22028734
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Onset Time of Mivacurium, Duration of Action of Mivacurium
MeSH Terms: interventions — Mivacurium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Butyrylcholinesterase activity determined by a blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elderly: patients aged 80 years or older
  Interventions: Drug: Mivacurium
- Young: patients aged 18-40 years
  Interventions: Drug: Mivacurium

INTERVENTIONS:
Drug: Mivacurium — 0.2 mg/kg based on ideal body weight calculated as height (cm) minus 105 for women and height (cm) minus 100 for men or actual body weight, whichever is lower
  Other Names: mivacron

SUMMARY:
The aim of this study is to determine the onset time, duration of action and effect on intubation conditions of mivacurium 0.2 mg/kg in elderly patients with age ≥ 80 years and in young patients aged 18 - 40 years.

DETAILED DESCRIPTION:
The aim of this study is to determine the onset time, duration of action and effect on intubation conditions of mivacurium 0.2 mg/kg in elderly patients with age ≥ 80 years and in young patients aged 18 - 40 years. The hypothesis of this study is that mivacurium administered in elderly patients (>80 years) has a longer onset time and duration of action compared to younger patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 80 or ≥ 18 to ≤ 40 years of age
2. Informed consent
3. Scheduled for elective surgery under general anaesthesia (expected duration of anaesthesia > 1 hour) with intubation and use of mivacurium
4. American Society of Anesthesiologists (ASA) physical status classification I to III
5. Can read and understand Danish

Exclusion Criteria:

1. Known allergy to mivacurium
2. Neuromuscular disease that may interfere with neuromuscular monitoring
3. Indication for rapid sequence induction
4. Surgery in the prone position
5. Known butyrylcholinesterase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients (≥ 80 years) and younger patients (18-40 years) scheduled for elective surgery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Onset time | within 10 minutes after administration of mivacurium
  the time from the start of the injection of mivacurium to train-of-four (TOF) count of 0 monitored by acceleromyography

SECONDARY OUTCOMES:
Duration of action | within 90 minutes after administration of mivacurium
  Duration of action is defined as time from start of mivacurium injection to reappearance of TOF ratio > 0.9.
Intubation conditions IDS | within 10 minutes after administration of mivacurium
  intubation conditions are rated according to intubating difficulty score IDS when TOF-ratio is 0.
Intubation conditions Fuchs-Buder | within 10 minutes after administration of mivacurium
  intubation conditions are rated according to Fuchs-Buder score when TOF-ratio is 0.
Laryngeal morbidity | 24 hours after surgery
  After 24 hours patients are asked about hoarseness and sore throat. Patients who experience either or both will be called 3 days postoperatively again. These two variables are assessed using a numeric ranking scale from 0 to 10.
Amount of ephedrine or metaoxedrine administered | within 10 minutes after administration of mivacurium
  If ephedrine or metaoxedrine is administered after induction of anaesthesia and until the patient is ready for properly positioning for surgery, it will be noted in the CRF, as well as the amount administered. Changes in blood pressure or heart rate are treated according to local guidelines.
Butyrylcholinesterase activity in a venous blood sample | within 7 days after administration of mivacurium
  Butyrylcholinesterase activity in a venous blood sample, and further determination of phenotype and genotype if the activity is low.

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, Principal Investigator — Rigshospitalet University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No